CLINICAL TRIAL: NCT00870922
Title: Effects of Masseter Manual Therapy on Temporomandibular Dysfunction: A Pilot Study
Brief Title: Effects of Masseter Manual Therapy on Temporomandibular Dysfunction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. James George, Jr, DC, Logan University, College of Chiropractic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR0204090171; 388
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Temporomandibular Joint; Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Disorder
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMD group (Experimental): Participants will receive ART and have Therabite (mouth opening) and pain (VAS) measured before and after ART
  Interventions: Procedure: Active release techniques

INTERVENTIONS:
Procedure: Active release techniques — Participants will receive ART and have Therabite (mouth opening) and pain (VAS) measured before and after ART

SUMMARY:
Muscles and myofascial dysfunction are more often the mechanism and source of pain in oral fascial disorders (OFD) than the TMJ. Masticatory muscles in patients with TMJ alterations are more hypertonic, less efficient and more prone to fatigue compared to age and sex matched controls. It is our opinion that Active Release Technique can be a reliable assessment and treatment tool in the resolution in cervical-cranio mandibular disorders. Our goal is to improve masticatory function through treatment of trigger points in the masseter.

DETAILED DESCRIPTION:
Recruit 45 patients with TMD determined by questionnaire. Measure pre and post mandibular active range of motion and VAS pain scale. Treatment will include 4 visits over a two week span measuring before first treatment and after last treatment. There will be 3 treatment groups; active release technique, post isometric relaxation and a no treatment control group. We will analyze data for any change in mandibular range of motion and VAS pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Difficulty and/or pain when opening mouth
* Jaw locking
* Difficulty or pain when chewing or talking
* TMJ clicking
* Jaw stiffness, tightness, or fatigue
* Pain in ear, temple or cheeks
* Frequent headaches, neckaches, toothaches
* Change in occlusion

Exclusion Criteria:

* Trauma to head, neck or jaw within last 12 months
* Recent dental extractions
* Taking prescription analgesics/muscle relaxants
* Recent cervical SMT (HVLA)
* Already under care for condition
* Sinus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 2 weeks

SECONDARY OUTCOMES:
VAS pain scale | 2 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States